A Study of Hookah Café Customers in the Atlanta Area

NCT05916170

IRB Approved Date: 08MAR2024

IRB00095123 Version Date: 12/4/2023

## A Study of Hookah Café Customers in the Atlanta Area Erin Sutfin, PhD, Principal Investigator

## INFORMED CONSENT FORM TO PARTICIPATE IN RESEARCH

You are eligible to participate in a study conducted by researchers at Wake Forest University School of Medicine in Winston-Salem, NC and Ewald and Wasserman Consulting, LLC. The purpose of this study is to understand the behavior and experiences of hookah café customers.

The study includes two phases. The first phase involves a brief survey and exhaling into a device so we can measure the particles in your breath. You will receive a \$25 electronic gift card for completing the first phase. After completing the first phase, you will enter the café as you had planned.

The second phase of the study will happen after you leave the café and will involve completing another brief survey and blowing into the tube we use to measure your breath particles. You will receive a \$50 electronic gift card for completing this phase.

Your participation is completely voluntary. You may stop participating at any time and you may skip any questions that you are not comfortable answering.

In this research study, any new information we collect from you about your health or behavior is considered Protected Health Information. We will make every effort to keep your Protected Health Information private. Your Protected Health Information will not be shared outside of our study team, and will be retained until the study is complete.

The risk of harm or discomfort that may happen as a result of taking part in this research study is not expected to be more than in daily life or from routine physical or psychological examinations or tests. There is a slight risk of breach of confidentiality; however, we will do our best to protect your confidential information.

You are not expected to receive any direct benefit from taking part in this research study. We hope the information learned from this study will benefit other people in the future. The alternative to participating in the study is to not participate.

| The person in charge of this study is Erin Suttin, PhD. If you have any questions, suggestions, or concerns | |
|---|---|
| regarding this study, or if you wish to withdraw from the study, please contact Dr. Sutfin at | |
| If you have any questions, suggestions, or concerns about your rights as | а |
| volunteer in this research, contact the Institutional Review Board at or the Research Subject | |
| Advocate at Wake Forest at | |